CLINICAL TRIAL: NCT04985942
Title: A Randomized, Double-Blind, Placebo-controlled Multicenter Study to Assess the Efficacy and Safety of Lumateperone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Brief Title: Clinical Trial of Lumateperone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITI-007-501
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Adjunctive MDD Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone 42 mg (Experimental)
  Interventions: Drug: Lumateperone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 42 mg capsules administered orally, once daily.
  Arms: Lumateperone 42 mg
Drug: Placebo — Matching capsules administered orally, once daily.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed-dose study in patients with a primary diagnosis of MDD according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) who have an inadequate response to ongoing ADT.

DETAILED DESCRIPTION:
The study will be conducted in three periods:

* Screening Period (up to 2 weeks) during which patient eligibility will be assessed;
* Double-blind Treatment Period (6 weeks) in which all patients will be randomized to receive placebo or lumateperone 42mg/day in 1:1 ratio.
* Safety Follow-up Period (1 week) in which all patients will return to the clinic for a safety follow-up visit approximately one week after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18 and 65 years, inclusive;
2. Meet DSM-5 diagnostic criteria for MDD (a diagnosis of MDD with psychotic features will be acceptable) as confirmed by the Investigator or Sponsor-approved rater using the Mini-International Neuropsychiatric Interview (MINI), and meet all the following criteria:

   1. The start of the current major depressive episode (MDE) is at least 8 weeks but not more than 18 months prior to Screening;
   2. Has at least moderate severity of illness based on rater-administered MADRS total score ≥ 24 at Screening and at Baseline;
   3. Has at least moderate severity of illness based on CGI-S score ≥ 4 at Screening and at Baseline;
   4. Has a Quick Inventory of Depressive Symptomatology-Self Report-16 item (QIDS-SR-16) score ≥14 at Screening and at Baseline;
   5. Has sufficient history and medical record confirmation verifying the ADT and the current MDE is causing clinically significant distress or impairment in social, occupational, or other important areas of functioning.
3. Currently having an inadequate response to ADT (less than 50% improvement) as confirmed by the Investigator and taking at least the minimum effective dose (per package insert) of one of the following antidepressants as monotherapy treatment for at least 6 weeks duration:

   1. citalopram/escitalopram
   2. fluoxetine
   3. paroxetine
   4. sertraline
   5. duloxetine
   6. levomilnacipran/milnacipran (if locally approved for MDD)
   7. venlafaxine/desvenlafaxine
   8. buproprion
   9. vilazodone
   10. vortioxetine

Exclusion Criteria:

1. Within the patient's lifetime, has a confirmed DSM-5 psychiatric diagnosis other than MDD, including:

   1. Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder or other psychotic disorder;
   2. Bipolar Disorder;
2. Within 6 months of Screening, has a confirmed DSM-5 psychiatric diagnosis other than MDD including:

   1. Anxiety disorders such as Panic Disorder or Generalized Anxiety Disorder; Obsessive-compulsive Disorder; Posttraumatic Stress Disorder as primary diagnoses.
   2. Eating disorder;
   3. Substance use disorders (excluding nicotine);
   4. Personality disorder of sufficient severity to have a major impact on the patient's psychiatric status;
   5. Within 12 months of Screening, has had any other psychiatric condition (other than MDD) that has been the main focus of treatment;
3. The patient experiences a ≥ 25% decrease in the MADRS total score between Screening and Baseline;
4. The patient experiences a ≥ 25% decrease in the QIDS-SR-16 total score between Screening and Baseline;
5. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during participation in the study or:

   1. At Screening, the patient scores "yes" on Suicidal Ideation Items 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) within 6 months prior to Screening, or at Baseline, the patient scores "yes" on Suicidal Ideation Items 4 or 5 since the Screening Visit;
   2. At Screening, the patient has had 1 or more suicide attempts within 2 years prior to Screening;
   3. At Screening or Baseline, the patient scores ≥ 5 on MADRS Item 10 (Suicidal Thoughts), or
   4. The patient is considered to be in imminent danger to him/herself or others.
6. The patient has a first MDE at age 60 years or older.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (15):
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Glendale, California
  - Clinical Site, Oceanside, California
  - Clinical Site, Redlands, California
  - Clinical Site, Temecula, California
  - Clinical Site, Upland, California
  - Clinical Site, Fort Lauderdale, Florida
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Berlin, New Jersey
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Cedarhurst, New York
  - Clinical Site, Austin, Texas
- Bulgaria (7):
  - Clinical Site, Burgas
  - Clinical Site, Kazanlak
  - Clinical Site, Pleven
  - Clinical Site, Rousse
  - Clinical Site, Tsarev Brod
  - Clinical Site, Veliko Tarnovo
  - Clinical Site, Vratsa
- Czechia (4):
  - Clinical Site, Brno
  - Clinical Site, Ostrava
  - Clinical site, Pilsen
  - Clinical Site, Prague
- Hungary (2):
  - Clinical Site, Budapest
  - Clinical Site, Gyöngyös
- India (14):
  - Clinical Site, Guwahati, Assam
  - Clinical Site, Ahmedabad, Gujarat
  - Clinical Site, Jūnāgadh, Gujarat
  - Clinical Site, Vadodara, Gujarat
  - Clinical Site, Mangaluru, Karnataka
  - Clinical Site, Mysore, Karnataka
  - Clinical Site, Kozhikode, Kerala
  - Clinical Site, Aurangabad, Maharashtra
  - Clinical Site, Nagpur, Maharashtra
  - Clinical Site, Nashik, Maharashtra
  - Clinical Site, Ludhiana, Punjab
  - Clinical Site, Jaipur, Rajasthan
  - Clinical Site, Lucknow, Uttar Pradesh
  - Clinical Site, Varanasi, Uttar Pradesh
- Slovakia (6):
  - Clinical Site, Bratislava
  - Clinical Site, Košice
  - Clinical Site, Rimavská Sobota
  - Clinical Site, Svidník
  - Clinical Site, Vranov nad Topľou
  - Clinical Site, Zlaté Moravce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durgam S, Earley WR, Kozauer SG, Chen C, Lakkis H, McIntyre RS, Stahl S. Lumateperone as Adjunctive Therapy in Patients With Major Depressive Disorder: Results From a Randomized, Double-Blind, Phase 3 Trial. J Clin Psychiatry. 2025 Aug 25;86(4):25m15848. doi: 10.4088/JCP.25m15848. PMID 40875502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumateperone 42 mg | Placebo
Started (485 patients were randomized; 484 patients received study drug and are included in the safety population.) | 241 | 243
Completed | 220 | 232
Not Completed | 21 | 11
Not completed — Adverse Event | 14 | 2
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumateperone 42 mg | Placebo | Total
Number analyzed (Participants) | 241 | 243 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.39) | 45.1 (12.51) | 45.0 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 160 | 318
  Male | 83 | 83 | 166
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 180 | 191 | 371
  Asian | 40 | 33 | 73
  Black or African American | 20 | 16 | 36
  Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Hungary | 6 | 10 | 16
  United States | 75 | 75 | 150
  Czechia | 51 | 54 | 105
  Slovakia | 21 | 18 | 39
  Bulgaria | 54 | 55 | 109
  India | 34 | 31 | 65
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
  units on a scale | 30.4 (3.76) | 30.0 (3.51) | 30.2 (3.64)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Åsberg Depression Rating Scale
Description: Change from baseline to Day 43 in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. The MADRS is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
Time Frame: Day 43
Population: The analysis of the primary and secondary efficacy outcome measures are based on the Modified Intent-to-Treat (mITT) Population which included 481 randomized patients. The mITT Population includes all randomized patients who received at least 1 dose of study drug, had a baseline MADRS total score, and who had at least one on-study drug, postbaseline MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42 mg | Placebo
Number analyzed (Participants) | 239 | 242
score on a scale | -14.7 (0.54) | -9.8 (0.53)
Statistical Analysis 1: Comparison: Lumateperone 42 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; MMRM Analysis Based on Hypothetical Estimand Strategy; Least Squares Mean Difference = -4.9, 95% CI 2-sided [-6.38 to -3.44], Standard Error of Mean 0.75

2. Secondary Outcome: Clinical Global Impression Scale-Severity
Description: Change from baseline to Day 43 in the Clinical Global Impression Scale-Severity (CGI-S). The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Day 43
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42 mg | Placebo
Number analyzed (Participants) | 239 | 242
score on a scale | -1.6 (0.07) | -0.9 (0.07)
Statistical Analysis 1: Comparison: Lumateperone 42 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; MMRM Analysis Based on Hypothetical Estimand Strategy; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.85 to -0.48], Standard Error of Mean 0.09

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~9 weeks), including 6 weeks of double-blind treatment.
Arm/Group | Lumateperone 42 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/243
Serious Adverse Events (participants affected / at risk) | 1/241 | 1/243
Other Adverse Events (participants affected / at risk) | 92/241 | 53/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumateperone 42 mg (N=241) | Placebo (N=243)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 42 mg (N=241) | Placebo (N=243)
Dry Mouth (Gastrointestinal disorders) | 26 | 5
Fatigue (General disorders) | 23 | 5
Tremor (Nervous system disorders) | 12 | 1
Headache (Nervous system disorders) | 38 | 37
Dizziness (Nervous system disorders) | 25 | 15
Nausea (Gastrointestinal disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04985942/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT04985942/SAP_001.pdf